CLINICAL TRIAL: NCT00077597
Title: A Randomized, Open-label Study of the Effect of Intravenous Mircera on Hemoglobin Level/Correction in Dialysis Patients With Chronic Kidney Disease
Brief Title: A Study of Mircera for the Treatment of Anemia in Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16736
Record Dates: First submitted 2004-02-10; First posted 2004-02-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Erythropoietin; continuous erythropoietin receptor activator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: epoetin

INTERVENTIONS:
Drug: epoetin — 3 times a week iv, as prescribed.
  Arms: 2
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 0.4 micrograms/kg iv (starting dose) once every 2 weeks
  Arms: 1

SUMMARY:
This study will assess the efficacy and safety of Mircera given intravenously in the treatment of renal anemia in chronic kidney disease patients on dialysis who are not currently receiving epoetin or any other erythropoietic substance. The anticipated time on study treatment is 1-2 years and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* chronic renal anemia;
* dialysis therapy for at least 2 weeks before screening.

Exclusion Criteria:

* women who are pregnant, breastfeeding or using unreliable birth control methods;
* administration of any investigational drug within 4 weeks before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2004-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Hemoglobin response rate | Weeks 1-24

SECONDARY OUTCOMES:
Hb over time, time to target Hb response, incidence of RBC transfusions. Vital signs, ECG, AEs, laboratory values\n | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (54):
- United States (14):
  - Davis, California
  - Lakewood, Colorado
  - Atlanta, Georgia
  - Augusta, Georgia
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Mineola, New York
  - New York, New York
  - Toledo, Ohio
  - Houston, Texas
  - Burlington, Vermont
  - Norfolk, Virginia
- Brazil (3):
  - Curitiba
  - Ribeirão Preto
  - São Paulo
- Canada (9):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Kingston, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Czechia (3):
  - Liberec
  - Prague
  - Ústí nad Labem
- Greece (4):
  - Alexandroupoli
  - Larissa
  - Nikaia
  - Thessaloniki
- Norway (2):
  - Bergen
  - Oslo
- Poland (8):
  - Gdansk
  - Gdynia
  - Krakow
  - Lodz
  - Poznan
  - Szczecin
  - Wołomin
  - Wroclaw
- Russia (2):
  - Moscow
  - Saint Petersburg
- South Africa (2):
  - Johannesburg
  - Soweto
- Spain (2):
  - Bilbao
  - Santander
- Karlstad, Sweden
- Lausanne, Switzerland
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Chon Buri

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Klinger M, Arias M, Vargemezis V, Besarab A, Sulowicz W, Gerntholtz T, Ciechanowski K, Dougherty FC, Beyer U. Efficacy of intravenous methoxy polyethylene glycol-epoetin beta administered every 2 weeks compared with epoetin administered 3 times weekly in patients treated by hemodialysis or peritoneal dialysis: a randomized trial. Am J Kidney Dis. 2007 Dec;50(6):989-1000. doi: 10.1053/j.ajkd.2007.08.013. PMID 18037099